CLINICAL TRIAL: NCT01631318
Title: Pilot Technical Feasibility Study on 3D Contrast-enhanced Ultrasound Imaging and to Assess Whether Change in Ultrasound 3D Perfusion Pattern Can Predict Treatment Response
Brief Title: Pilot 3D Contrast-Enhanced Ultrasound Imaging to Predict Treatment Response in Liver Metastases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-24334; NCI-2012-01008 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 1R01CA195443 (NIH); HEP0043 (Other: OnCore)
Record Dates: First submitted 2012-06-26; First posted 2012-06-29 (Estimated); Last update posted 2022-06-10 (Actual); Status verified 2022-06

CONDITIONS: Liver Metastases; Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (3D contrast-enhanced ultrasound imaging) (Experimental): Patients undergo 3D dynamic contrast-enhanced ultrasound imaging before initiation of chemotherapy and at 2 weeks.
  Interventions: Procedure: Dynamic contrast-enhanced ultrasound imaging; Device: Optical Tracking Device; Device: Electromagnetic Tracking Device; Drug: Perflutren

INTERVENTIONS:
Procedure: Dynamic contrast-enhanced ultrasound imaging — Ultrasound imaging procedure
  Other Names: DCE-USI; 3D contrast enhanced ultrasound imaging
Device: Optical Tracking Device — Optical Tracking Device, manufactured by Atracsys LLC, Switzerland.
Device: Electromagnetic Tracking Device — Electromagnetic Tracking Device, Ascension Technology Corporation, Milton, Vermont.
Drug: Perflutren — Perflutren lipid microsphere, IV 0.4 mL. Used as standard contrast agent, not the subject of the study.
  Other Names: Definity

SUMMARY:
Patients are invited to participate in a research study of liver perfusion (how blood flows to the liver over time). Researchers hope to learn whether perfusion characteristics of liver metastases may be predictive of response to treatment and whether liver perfusion characteristics can be used to follow response to treatment. Patients were selected as a possible participant in this study because they are identified as having liver metastases

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The purpose of this study is to perform a pilot feasibility study on 3-dimensional (3D) ultrasound imaging of liver metastases and to evaluate whether perfusion characteristics (measurements of blood-flow) of hepatic metastases can predict tumor response to treatment in patients with liver metastases. The investigators long term goal is to assess whether early perfusion changes at 2 weeks after chemotherapy initiation can be used as a non-invasive early biomarker for treatment response assessment.

OUTLINE:

Patients undergo 3D dynamic contrast-enhanced ultrasound imaging before initiation of chemotherapy, at 2 weeks, and at 2 months.

ELIGIBILITY:
Inclusion Criteria

* Provides written Informed Consent and is willing to comply with protocol requirements.
* Has at least 1 focal lesion in liver or kidney
* Patient may be (i) in the process of receiving treatment (1 scan session), (ii) never treated (3 scan sessions) or (iii) changing treatment regimen/ type and/or receiving a new form of treatment and/or has been on a treatment break ('holiday')(3 scan session)
* Is at least18 years of age.

Exclusion Criteria

* Is determined by the Investigator that the subject is clinically unsuitable for the study.
* Known right to left cardiac shunt, bidirectional or transient.
* Hypersensitivity to perflutren.
* Hypersenstivity to the contrast agent Definity.
* Pregnant and lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-11-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Measurements of blood flow, in terms of comparison of the perfusion parameters of the lesion as a predictor of tumor response to treatment and use as a biomarker for response to treatment | Baseline
  Descriptive statistics will be presented for lesion size, by lesion type, and across lesion types. Lesion shape, depth, vascularization, and border definition will also be categorized by dose and lesion type. Based on the unenhanced ultrasound, the target lesion to liver echogenicity will be categorized by lesion type. Based on the Definity®-enhanced ultrasound, the pattern of enhancement of the target lesion will be summarized by lesion type.
Measurements of blood flow, in terms of comparison of the perfusion parameters of the lesion as a predictor of tumor response to treatment and use as a biomarker for response to treatment | 2 weeks after chemotherapy initiation
  Descriptive statistics will be presented for lesion size, by lesion type, and across lesion types. Lesion shape, depth, vascularization, and border definition will also be categorized by dose and lesion type. Based on the unenhanced ultrasound, the target lesion to liver echogenicity will be categorized by lesion type. Based on the Definity®-enhanced ultrasound, the pattern of enhancement of the target lesion will be summarized by lesion type.
Measurements of blood flow, in terms of comparison of the perfusion parameters of the lesion as a predictor of tumor response to treatment and use as a biomarker for response to treatment | 2 months post-treatment
  Descriptive statistics will be presented for lesion size, by lesion type, and across lesion types. Lesion shape, depth, vascularization, and border definition will also be categorized by dose and lesion type. Based on the unenhanced ultrasound, the target lesion to liver echogenicity will be categorized by lesion type. Based on the Definity®-enhanced ultrasound, the pattern of enhancement of the target lesion will be summarized by lesion type.

CONTACTS AND LOCATIONS:
Overall Officials: Aya Kamaya, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No